CLINICAL TRIAL: NCT00414752
Title: A Randomized, Double Blind, Multiple Dose, Cross-Over, Placebo- and Active-Controlled Proof of Concept Study to Explore the Effects of AFQ056 and Nicotine (Active Comparator) on Craving and Withdrawal During Voluntary Smoking Abstinence in Healthy Smokers
Brief Title: Effects of AFQ056 and Nicotine in Reducing Cigarette Smoking
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAFQ056A2109
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Smoking Abstinence
Keywords: Smoking, abstinence, craving, smoker, AFQ056, nicotine, placebo
MeSH Terms: conditions — Smoking

INTERVENTIONS:
Drug: AFQ065

SUMMARY:
The purpose of this study is to assess the safety and efficacy of AFQ056 and nicotine compared to placebo on craving and withdrawal symptoms during voluntary smoking stoppage in healthy smokers. This study will also assess how the body interacts with AFQ056.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male & female subjects at least 18 years and ≤60 years of age
* In good health
* Female subjects must be surgically sterilized or postmenopausal.
* Current smokers not intending to quit
* Smoke on average 15 cigarettes or more and less than 60 cigarettes a day for the past year
* Fagerström Test for Nicotine Dependence score of at least 5 (indicates moderate to heavy smokers)
* Willing to refrain from smoking as required
* Written informed consent before entering the study

Exclusion Criteria:

* History of heart disease, septum defect and/or cardiac valves surgery; clinical relevant abnormality in the ECG
* Investigational drug treatment within 4 weeks prior to screening unless local health authority guidelines mandate a longer period
* Women of childbearing potential, pregnant or lactating females
* Donation of one unit (400mL) or more of blood, significant blood loss equaling at least one unit of blood within the past 2 months or a blood transfusion within 8 weeks prior to screening.
* Coffee consumption of more than 6 cups coffee/day
* Use of a medication within 2 weeks prior to Day 1 of each treatment period

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2006-09

PRIMARY OUTCOMES:
Reduction of craving by self-report questionnaires during 3 days of voluntary smoking stoppage

SECONDARY OUTCOMES:
Reduction in symptoms of withdrawal during 3 days of voluntary smoking stoppage
Reduction in nicotine consumption during 6 days of free smoking
Reduction in impulsivity during 3 days of free smoking and during 3 days of voluntary smoking stoppage
Reduction in craving during 6 days of free smoking
Safety and tolerability of AFQ056 during treatment periods
Assessment of how the body interacts with AFQ056

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Nuremberg, Germany